CLINICAL TRIAL: NCT02359279
Title: Radiographic Contrast To Differentiate Cavitated From Non-cavitated Tooth Decay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Principal Investigator, Douglas K Benn DDS, PhD, Principal Investigator, Creighton University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2R42DE023003-02 (NIH)
Record Dates: First submitted 2015-02-02; First posted 2015-02-10 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Contrast (Experimental): All subjects will be in one group who will have a control radiograph before applying sodium iodide to interproximal surfaces of teeth when another radiograph will be taken to test for the presence of caries cavitation.
  Interventions: Device: Sodium iodide

INTERVENTIONS:
Device: Sodium iodide — Comparison of control radiographs made before application of sodium iodide and test radiograph after application.

SUMMARY:
The proposed test is intended to enable dentists to differentiate between cavitated and non-cavitated tooth decay in the areas where teeth are in contact (interproximal surfaces). In these areas, dentists cannot visually inspect for caries, and currently bitewing X-rays (BWs) only correctly detect the presence of enamel decay 15-25% of the time. This low sensitivity can lead to late treatment resulting in unnecessarily large fillings, crowns, pain, root canals, and possible later loss of teeth.

DETAILED DESCRIPTION:
Tooth sites will be recorded by both tooth number, type of surface (mesial, distal, occlusal), cavitated, non-cavitated, healthy. Radiographs will similarly be scored. Although contrast agents are classified as drugs this is not a study of drug properties or effect on cells since the properties of the agent are already well known and its safety record well established. This study will be recording the radiopacity of the contrast agent on healthy tooth surfaces, non-cavitated tooth surfaces and cavitated tooth surfaces. The outcome for each surface type will be presence or absence of a radiopacity on a radiograph which will be made at the one and only visit for each study subject. The radiograph contains the data from the intervention (placement of contrast agent) and the outcome will be assessed some weeks later after the completion of the data collection.

ELIGIBILITY:
Inclusion Criteria:

* Must have a minimum of 2 adjacent teeth so that interproximal surfaces of interest are in contact and hidden from direct visual examination.

The occlusal plane plane should be normal so that the interproximal contact regions are normal.

English or Spanish speaker.

Exclusion Criteria:

* Pregnant women. A person who has participated in a similar study involving dental radiography within the last 12 months.

Fillings must not be present in the regions of interest.

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of cavitated versus non-cavitated caries lesions in 116 tooth surfaces. | Immediately after application of sodium iodide
  The PI will perform the clinical application of the sodium iodide and radiograph the subject. A control radiograph will be taken of tooth crowns before the application of the contrast. Immediately after the contrast application another radiograph will be exposed. If caries is present a lucency will be seen in the control The test radiograph will show either contrast on the tooth surface (non-cavitated) or below the surface (caviiatetd). Rubber impressions will be made of the tooth surfaces and scanned with a laser to provide a 3D replica which will be the gold standard for presence or absence of cavitation. At a later date 3 independent dentists will be provided with blinded radiographs in a randomized order to report the presence or absence of cavitated cries lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Benn, DDS PhD, Principal Investigator — Creighton University & Firefly Health Innovations NE inc
Locations (1):
- Creighton University School of Dentistry, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benn DK, Cooper RL, Nunn ME, Edwards SE, Rocha-Sanchez SM. A radiographic method for distinguishing noncavitated from cavitated proximal carious lesions: A proof of concept clinical trial. Oral Surg Oral Med Oral Pathol Oral Radiol. 2021 Dec;132(6):715-726. doi: 10.1016/j.oooo.2021.02.014. Epub 2021 Feb 23. PMID 34083157